CLINICAL TRIAL: NCT01347008
Title: Effect of Sildenafil on the Microcirculatory Blood Flow and on the Endothelial Progenitor Cells in Patients With Systemic Sclerosis: a Randomized, Double-blind, Placebo-controlled Clinical Trial
Brief Title: Effect of Sildenafil on the Microcirculatory Blood Flow and Endothelial Progenitor Cells in Systemic Sclerosis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Federal University of São Paulo (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Principal Investigator, Fernando Villela Andrigueti, MD, Federal University of São Paulo
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FAPESP 2011/00012-3
Record Dates: First submitted 2011-05-02; First posted 2011-05-04 (Estimated); Results first posted 2016-12-05 (Estimated); Last update posted 2016-12-05 (Estimated); Status verified 2016-10

CONDITIONS: Scleroderma, Systemic; Scleroderma, Diffuse; Scleroderma, Limited; Raynaud Phenomenon
Keywords: Sildenafil; Endothelial Progenitor Cells; Laser Doppler Imaging
MeSH Terms: conditions — Scleroderma, Systemic; Scleroderma, Diffuse; Scleroderma, Limited; Raynaud Disease | interventions — Sildenafil Citrate; Long-Term Synaptic Depression; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sildenafil citrate (Active Comparator): Oral Sildenafil citrate, 50mg, b.i.d.
  Interventions: Drug: Sildenafil citrate
- Sugar pill (Placebo Comparator): Placebo pill (identical to Sildenafil citrate 50mg), b.i.d.
  Interventions: Drug: Placebo (Sugar pill)

INTERVENTIONS:
Drug: Sildenafil citrate — Oral sildenafil citratre, 50mg b.i.d., 8 weeks
  Other Names: Sildenafil citrate, EMS Sigma Pharma, Ltd, Brazil
  Arms: Sildenafil citrate
Drug: Placebo (Sugar pill) — Placebo pills similar to sildenafil citrate pills, b.i.d for 8 weeks
  Other Names: Placebo
  Arms: Sugar pill

SUMMARY:
Early phases of systemic sclerosis is characterized by inflammatory and microvasculature alterations. Sildenafil citrate has been shown to have vasodilatory effects and to enhance vasculogenesis. The purpose of this study is to evaluate the effect of sildenafil citrate on hand blood flow of patients with systemic sclerosis, using Laser Doppler Imaging.

DETAILED DESCRIPTION:
Progressive microangiopathy and endothelial dysfunction are identified in early phases of systemic sclerosis. These alterations may result in progressive reduction of vessel lumen, decreased blood flow, and a state of chronic hypoxia resulting in digital ulcers, digital pitting, and, in more severe cases, gangrene and amputation of the extremities. Few studies aimed to evaluate the effects of Sildenafil on the microcirculatory blood flow in patients with Raynaud's phenomenon secondary to systemic sclerosis (SS). Moreover, no study has evaluated the effect of this drug on the number and function of endothelial progenitor cells in SS patients. The relatively new technique of laser Doppler imaging (LDI) allows an objective measurement of superficial cutaneous microvascular blood flow and constitutes a promising approach in the assessment of the digital microvascular vasoreactivity in response to cold stimulus or in response to treatment in SSc patients.

ELIGIBILITY:
Inclusion Criteria:

* Systemic sclerosis according to the classification criteria of the American College of Rheumatology (1980) with no more than 4 years since diagnosis
* Early systemic sclerosis as defined by LeRoy and Medsger (2001)
* 6 or more Raynaud's crisis per week
* Written informed consent provided by the subjects prior to initiating study procedures

Exclusion Criteria:

* Smoking
* Peripheral or central vasculopathy other than Systemic sclerosis
* Uncontrolled Diabetes
* Liver disease
* Pregnant or lactating woman
* Current use of cyclosporin, prostanoids, bosentan or any PDE-5 inhibitors (including current Sildenafil use during randomization)
* History of stroke, myocardial infarction or life threatening cardiac condition within the last 6 months
* History of surgical sympathectomy
* Systolic blood pressure < 85mm Hg
* History of scleroderma renal crisis
* Known hypersensitivity to Sildenafil or any of the excipients
* History of Retinitis Pigmentosa
* Current use of Nitrates

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2011-04; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Fernando V Andrigueti, MD, Principal Investigator — Federal University of São Paulo
Locations (1):
- Systemic Sclerosis Outpatient Clinic, Hospital Sao Paulo, UNIFESP, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Maltez N, Maxwell LJ, Rirash F, Tanjong Ghogomu E, Harding SE, Tingey PC, Wells GA, Tugwell P, Pope J. Phosphodiesterase 5 inhibitors (PDE5i) for the treatment of Raynaud's phenomenon. Cochrane Database Syst Rev. 2023 Nov 6;11(11):CD014089. doi: 10.1002/14651858.CD014089. PMID 37929840

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients recruited at the Outpatient Clinic of The Federal University of Sao Paulo, between August 2011 and November 2012
Groups:
- Sugar Pill: Placebo: Placebo pills similar to sildenafil citrate pills, b.i.d for 8 weeks
Period: Overall Study
Arm/Group | Sildenafil Citrate | Sugar Pill
Started | 21 | 20
Completed | 21 | 20
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sildenafil Citrate | Sugar Pill | Total
Number analyzed (Participants) | 21 | 20 | 41
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.2 (10.9) | 41.6 (13.3) | 44.5 (12.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 20 | 41
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Brazil | 21 | 20 | 41
Digital skin microvascular blood flow measured by Laser Doppler Imaging (LDI) before cold stimulus [Mean (Standard Deviation); unit: perfusion units] — Finger blood flow of the four medial fingers, measured by laser Doppler imaging and expressed in arbitrary perfusion units (p.u.).
  perfusion units | 213.1 (87.9) | 241.9 (104.4) | 234.6 (105.8)
Digital skin microvascular blood flow measured by Laser Doppler Imaging (LDI) after cold stimulus. [Mean (Standard Deviation); unit: perfusion units] — Finger blood flow of the four medial fingers, measured by laser Doppler imaging and expressed in arbitrary perfusion units (p.u.). Measure taken after submersion of both hands in water at 15°C for 1 minute.
  perfusion units | 178.8 (92.4) | 218.6 (98.9) | 200.2 (96.1)
Daily frequency of Raynuad's Phenomenon attacks [Mean (Standard Deviation); unit: number of attacks per day] — Daily frequency of RP attacks as self registered in a 1-week diary. Any episode of pallor or cyanosis of the hand/fingers was considered as a RP attack, and patients were supposed to register the daily amount of such episodes on a 1-week diary, previously to the medical visit.
  number of attacks per day | 2.3 (2.5) | 1.9 (2.0) | 2.1 (2.3)

OUTCOME MEASURES:

1. Primary Outcome: Digital Skin Microvascular Blood Flow Measured by Laser Doppler Imaging (LDI) Before Cold Stimulus
Description: Finger blood flow of the four medial fingers, measured by laser Doppler imaging and expressed in arbitrary perfusion units (p.u.).
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: perfusion units
Arm/Group | Sildenafil Citrate | Sugar Pill
Number analyzed (Participants) | 21 | 20
perfusion units | 260.0 (108.0) | 246.3 (122.6)

2. Primary Outcome: Digital Skin Microvascular Blood Flow Measured by Laser Doppler Imaging (LDI) After Cold Stimulus.
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: perfusion units
Arm/Group | Sildenafil Citrate | Sugar Pill
Number analyzed (Participants) | 21 | 20
perfusion units | 257.7 (123.3) | 220.5 (119.9)

3. Secondary Outcome: Daily Frequency of Raynaud's Phenomenon Attacks
Description: Daily frequency of RP attacks as self registered in a 1-week diary. Any episode of pallor or cyanosis of the hand/fingers was considered as a RP attack, and patients were supposed to register the daily amount of such episodes on a 1-week diary, previously to the medical visit.
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: number of attacks per day
Arm/Group | Sildenafil Citrate | Sugar Pill
Number analyzed (Participants) | 21 | 20
number of attacks per day | 1.9 (2.4) | 1.7 (2.2)

ADVERSE EVENTS:
Time Frame: 10 weeks
Arm/Group | Sildenafil Citrate | Sugar Pill
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/20
Other Adverse Events (participants affected / at risk) | 7/21 | 1/20
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Sildenafil Citrate (N=21) | Sugar Pill (N=20)
Headache (Nervous system disorders) | 7 | 1

LIMITATIONS AND CAVEATS:
Small numbers of subjects analyzed; blood flow differences due to outside temperature variations

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No